CLINICAL TRIAL: NCT07166640
Title: Estimation of the Median Effective Dose of Propofol for Colonoscope Insertion in Adult Patients: A Prospective Dose-Finding Study
Brief Title: Propofol Dose-Finding for Colonoscope Insertion in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Bedirhan Günel, Principal Investigator, Kocaeli City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSH-ANREA-BG-07
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group mono-Propofol (Other): The study is designed using Dixon's up-and-down sequential allocation method. Successful colonoscope insertion is defined as the absence of pain, movement, or vocal response, together with a MOAA/S score ≤2 at the second minute after induction, and maintained until the colonoscope passes the rectosigmoid junction. In cases of failure, an additional dose of propofol is administered, and the initial dose for the next patient is increased by 0.1 mg/kg. In cases of success, the initial dose for the next patient is decreased by 0.1 mg/kg.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — The initial dose is 1.5 mg/kg, adjusted in increments or decrements of 0.1 mg/kg according to the modified Dixon's up-and-down method. Additional rescue doses of 0.25-0.5 mg/kg is titrated if insertion is unsuccessful.

SUMMARY:
The aim of this prospective dose-finding study is to determine the ED50 of propofol required for successful colonoscope insertion in adult patients. The study is designed using Dixon's up-and-down sequential allocation method. Successful colonoscope insertion is defined as the absence of pain, movement, or vocal response, together with a MOAA/S score ≤2 at the second minute after induction, and maintained until the colonoscope passes the rectosigmoid junction. In cases of failure, an additional dose of propofol is administered, and the initial dose for the next patient is increased by 0.1 mg/kg. In cases of success, the initial dose for the next patient is decreased by 0.1 mg/kg.

The primary outcome is the determination of the ED50 of propofol for successful colonoscope insertion until passage of the rectosigmoid junction.

DETAILED DESCRIPTION:
The procedure is performed by an experienced endoscopist. If, during passage of the colonoscope through the rectosigmoid junction, the patient moves, experiences pain, vocalizes, or if the MOAA/S score is ≥3 at the second minute after induction, the insertion is defined as unsuccessful, and an additional rescue dose of 0.25-0.5 mg/kg propofol is titrated intravenously. The initial propofol dose for the next patient is then increased by 0.1 mg/kg.

If there is no movement during passage of the rectosigmoid junction, the patient reports no pain, and the MOAA/S score is ≤2 at the second minute after induction, the insertion is defined as successful, and the initial dose for the next patient is decreased by 0.1 mg/kg.

The conditions for colonoscope insertion are evaluated only at the initial attempt. If, after the start of the procedure, the patient experiences pain, moves, vocalizes, or the MOAA/S score is ≥3, an additional dose of 0.25-0.5 mg/kg propofol is titrated as required.

Throughout the procedure, the target is to maintain a MOAA/S score ≤2, which is systematically assessed at 2-minute intervals. Vital signs, procedure duration, and drug dosages are recorded for all patients.

At the end of the procedure, patients are awakened with verbal and tactile stimuli. After completion of colonoscopy, all patients are transferred to the post-anesthesia care unit for close monitoring until achieving a Modified Aldrete score of 10. Patients with a Modified Aldrete score of 10 are discharged.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provided informed consent to participate
* Patients scheduled for colonoscopy
* ASA physical status I-III
* Male and female patients aged 18-65 years

Exclusion Criteria:

* Patients who did not provide consent
* Known allergy to propofol
* Body weight <40 kg
* Body mass index (BMI) >30 kg/m²
* Presence of acute or chronic pain
* Chronic alcohol consumption
* Use of antipsychotic, antidepressant, or hypnotic medications
* Patients with obstructive sleep apnea syndrome (STOP-Bang score ≥3)
* Patients with known anorectal diseases such as hemorrhoids, anal fissure, or anal fistula
* History of oncological disease
* Uncontrolled hypertension (blood pressure >180/110 mmHg)
* Severe hepatic or renal dysfunction
* Acute respiratory tract infection or other chronic respiratory disorders
* Patients with a history of colorectal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
ED50 | At 2 minutes after induction (during colonoscope insertion)
  The median effective dose (ED50) of propofol required for successful colonoscope insertion in geriatric patients will be determined using the modified Dixon's up-and-down method. Successful insertion is defined as the absence of movement or vocalization and a MOAA/S score ≤2 within 2 minutes after induction, maintained until the colonoscope passes the rectosigmoid junction.

SECONDARY OUTCOMES:
ED95 | At 2 minutes after induction (during colonoscope insertion)
  The median effective dose (ED95) of propofol required for successful colonoscope insertion in geriatric patients will be determined using the modified Dixon's up-and-down method. Successful insertion is defined as the absence of movement or vocalization and a MOAA/S score ≤2 within 2 minutes after induction, maintained until the colonoscope passes the rectosigmoid junction.
Additional propofol dose | The cumulative amount of rescue propofol administered during the procedure will be recorded.
  After induction until the end of the colonoscopy procedure
total propofol dose | The cumulative amount of total propofol administered during the procedure will be recorded.
  From induction until the end of the colonoscopy procedure
Presence of pain during propofol injection | Immediately after first propofol administration
  Pain during propofol injection will be assessed as a binary variable (Yes/No), evaluated immediately after the first propofol injection. Presence of pain = Yes, Absence of pain = No.
Heart rate | Baseline (before sedation); at colonoscope insertion (start of procedure); 2 minutes after insertion; and at the end of the procedure (completion of colonoscopy).
  Hemodynamic parameters will be recorded at the specified time points to evaluate physiological stability during the procedure.
mean arterial pressure | Baseline (before sedation); at colonoscope insertion (start of procedure); 2 minutes after insertion; and at the end of the procedure (completion of colonoscopy).
  Hemodynamic parameters will be recorded at the specified time points to evaluate physiological stability during the procedure.
SpO2 | Baseline (before sedation); at colonoscope insertion (start of procedure); 2 minutes after insertion; and at the end of the procedure (completion of colonoscopy).
  oxygen saturation parameter will be recorded at the specified time points to evaluate physiological stability during the procedure.
Procedure interruptions due to airway interventions | Throughout the colonoscopy procedure
  The incidence of airway interventions (chin lift, jaw thrust, mask ventilation) and associated procedural interruptions will be recorded.
Minimum SpO₂ value during the procedure | Throughout the colonoscopy procedure
  The lowest SpO₂ value observed during the procedure will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Bedirhan Günel, Principal Investigator — Kocaeli City Hospital
Locations (1):
- University of Health Sciences Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu FK, Wan L, Shao LJZ, Zou Y, Liu SH, Xue FS. Estimation of effective dose of propofol mono-sedation for successful insertion of upper gastrointestinal endoscope in healthy, non-obese Chinese adults. J Clin Pharm Ther. 2021 Apr;46(2):484-491. doi: 10.1111/jcpt.13312. Epub 2020 Nov 20. PMID 33217028